CLINICAL TRIAL: NCT00263367
Title: Effect of Hyperbaric Therapy on Markers of Oxidative Stress in Children With Autism: A Pilot Study
Brief Title: Effect of Hyperbaric Therapy on Markers of Oxidative Stress in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The International Child Development Resource Center (Other)
Responsible Party: James Bradstreet MD, ICDRC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICDRC-22.2005
Record Dates: First submitted 2005-11-21; First posted 2005-12-08 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Autism; Oxidative Stress
Keywords: Autism; Oxidative Stress; Hyperbaric Oxygen; Reduced Glutathione; Lipid Peroxides
MeSH Terms: conditions — Autistic Disorder | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hyperbaric oxygen at 1.3 ATA (Other): Hyperbaric Oxygen at 1.3 ATA for one hour followed by measurement of glutathione in the blood
  Interventions: Other: Hyperbaric Oxygen

INTERVENTIONS:
Other: Hyperbaric Oxygen — Hyperbaric Oxygen at 1.3 ATA for one hour
  Other Names: HBOT

SUMMARY:
This study will look at the changes taking place in the blood levels of key markers of oxidative stress. Oxidative stress is the biological equivalent of rust on a car. It changes vital cell chemistry. It is known to occur at high pressure oxygen, but little is known about changes at pressures slightly greater than normal atmospheric pressure.

Hyperbaric therapy is used in a variety of medical conditions. It is being tested in this study only for safety. It is not being assessed for the ability of hyperbaric oxygen to improve the clinical condition of children with autism.

This study was felt to be important since autism appears to be associated with oxidative stress and hyperbarics was being used "off-label" for this condition without safety studies.

DETAILED DESCRIPTION:
Blood will be drawn immediately prior to a one hour session of hyperbarics (HBT. A catheter will be inserted in to a vein and converted to a heparin lock indwelling port for the next blood draw. The child (ages 5-12 years) will then undergo 1 hour of compression at 1.3 atmospheric pressure (4 psi above room air pressure). Supplemental oxygen will be provided to the child.

A second blood draw from the catheter site will be accomplished immediately after the child comes out of the HBT chamber.

These will be sent to the laboratories for evaluation of changes in reduced glutathione and lipid peroxides.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with autism ages 5-12 and undergoing hyperbarics

Exclusion Criteria:

* Seizures, acute URI, or inability to ventilate ears

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2005-10; Primary Completion 2006-01 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
glutathione | 1 hour
  measurement of glutathione immediately after one hour of exposure to low dose HBOT

CONTACTS AND LOCATIONS:
Overall Officials: James J Bradstreet, MD FAAFP, Principal Investigator — ICDRC
Locations (1):
- ICDRC, Melbourne, Florida, United States

REFERENCES:
- See also: Primary Location — http://icdrc.org